CLINICAL TRIAL: NCT03405844
Title: The Effectiveness of a Static Passive Stretching on Glenohumeral Rotation Range of Movement in Elite Swimmers After Competition: A Quasi-experimental Clinical Trial
Brief Title: A Static Passive Stretching on Glenohumeral Rotation Range of Movement in Elite Swimmers
Status: Completed | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Jorge Hugo Villafañe, PhD, Researcher, Fondazione Don Carlo Gnocchi Onlus
Other Study IDs: SETRADE
Record Dates: First submitted 2018-01-15; First posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Shoulder Injury
Keywords: Shoulder; glenohumeral; stretching
MeSH Terms: conditions — Shoulder Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Shoulder injury is a common problem of overhead athletes, as swimmers. It's reported a reduction of side-to-side glenohumeral rotation from 11 to 18 degrees can increase 1.9 points the injury risk, because an alteration in biomechanics can turn lead to clinical findings of impingement and labral pathology. Posterior deltoid is a main muscle for propulsion in swimming stroke. To our knowledge, it isn't known how a posterior deltoid static passive stretch could reduce glenohumeral rotation restriction after swimming competition.

ELIGIBILITY:
Inclusion Criteria:

* elite swimmers

Exclusion Criteria:

* shoulder surgery
* dislocation

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Swimmers from the winter national trials who competed at state, national or international level, performed at least five swim sessions per week and intended to continue this training level during the following 24 months were eligible to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
Change of glenohumeral rotation degrees | Basline
  Internal and external rotation range of movement

CONTACTS AND LOCATIONS:
Overall Officials: JORGE H VILLAFAÑE, PhD, Principal Investigator — IRCCS Don Gnocchi Foundation
Locations (1):
- Jorge Hugo Villafañe, Milan, Italy

IPD SHARING:
Plan to Share IPD: No